CLINICAL TRIAL: NCT03617276
Title: A Study Investigating the Inter- and Intra- Rater Reliability of Functional Outcome Measures in Neurofibromatosis 2
Brief Title: Reliability of Functional Outcome Measures in Neurofibromatosis 2
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 16/NW/0504
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Neurofibromatosis 2
MeSH Terms: conditions — Neurofibromatosis 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outcome measurement: Each participant will be asked to complete each standardised outcome measure (SOM) three times and each trial will be videotaped by the researcher. The selected SOM's are the modified nine-hole peg test, the four square step test and the modified clinical test of sensory integration and balance. A doctor will watch the video on 2 separate occasions to evaluate intra-rater reliability. Inter-rater reliability will be assessed through asking three other neurofibromatosis specialist professionals (two NF2 consultants and one NF2 specialist nurse) to review the video and to score each measure completed. Once the filmed sessions have been analysed by the relevant clinician's the data will be destroyed in line with Trust policy. Each participant will also be required to complete the INFI-QOL questionnaire, the dynamic visual acuity test and provide information about the number of falls/near misses they have had over the past 12 months

SUMMARY:
Neurofibromatosis 2 (NF2) is a rare inherited condition. Those with NF2 usually present with tumours (schwannomas) in their inner ear, or vestibular organ, with common symptoms including problems with hearing, balance, dizziness and vision. This study aims to evaluate the reliability (stability) of a range of functional standardised outcome measures in adults with NF2.

DETAILED DESCRIPTION:
Neurofibromatosis 2 (NF2) is an inherited condition that occurs in 1 in 33,000 births; affecting hearing, balance, dizziness and vision primarily related to tumours (schwannomas) in the inner ear or other tumours which develop within the central nervous system. Neuropathy may also be an issue for people with NF2.

The complications of NF2 can lead to varied difficulties with activities of daily living and may impair quality of life. More recently, new pharmacological treatments for NF2 are being trialed which may have the potential to dramatically influence quality of life for people with NF2. Currently, evaluation of treatment effect in NF2 is based on a clinician's neurological assessment and imaging. However, imaging results do not always correlate with clinical and reported functional changes of the individual. Therefore, evaluating the effect of interventions or treatment should include the evaluation of a person's function using standardised outcome measures. The findings from this study will improve the care of people with NF2 by ensuring that we are able to measure functional changes in a person with NF2 with greater confidence, meaning that we can start, continue or cease treatments based on the holistic picture of an individual.

The world confederation of physiotherapists (WCPT) stipulates that standardised outcome measures (SOM) are used to provide a quantitative measure of capability, and to evaluate the impact of treatment on function. There are a wide range of SOM's that evaluate function so a SOM is chosen by the clinician based on the patient's presenting functional difficulty and the scientific credibility of the SOM. Scientific credibility (robustness) is based on scientific properties of the SOM i.e. how stable the SOM is (reliability) and whether it assesses what it is intending to assess (validity). It is important to evaluate each SOM within the target population as variability within that condition, strongly influences the SOM's reliability and validity (de Vel 2011).

At present, functional SOM's have limited scientific and subsequent clinical credibility when used in people with NF2 because their scientific properties have not yet been evaluated within this patient group which means that if they are used clinically or within research, there is an inherent element of doubt when interpreting the SOM's results. The objective of this research team is to create a core set of functional SOM's which have undergone rigorous scientific evaluation so that they can be used in the future for clinical practice and for research purposes in adults with NF2.

This study primarily aims to evaluate three commonly used SOM's for reliability in adults with NF2 (over 16 years of age). The measures chosen for evaluation are the nine hole peg test, the four square step test and the modified clinical test of sensory integration and balance (mCTSIB). Interrater reliability (the test result remains the same when reviewed by different people) and intrarater reliability (the test result remains stable when reviewed twice by the same tester) will be evaluated. From this data, we will be able to calculate the standard error of measurement an additional important scientific characteristics of SOM evaluation. A secondary objective is to correlate SOM objective markers with a subjective disease specific quality of life measure (NFTI-QOL) and self-reported falls rate and near misses. We will also collect data on dynamic visual acuity in this patient group.

ELIGIBILITY:
Inclusion Criteria:

Fulfill diagnostic criteria for NF2 Aged 16 years or older Attend the national NF service at Guys and St Thomas' NHS Foundation Trust Are able to provide informed consent Do not have any non-NF2 related comorbidities that affect mobility or balance (confirmed by the treating clinician) Are able to walk more than 10m without assistance of a person Do not have unstable vascular or orthopaedic pathology at the cervical spine (confirmed by consultant) Have not had a stroke within the last 3 months

Exclusion Criteria:

Do not fulfill diagnostic criteria for NF2 Aged under 16 years or older Are unable to provide informed consent Have non-NF2 related comorbidities that affect mobility or balance (confirmed by the treating clinician) Are unable to walk more than 10m without assistance of a person Have unstable vascular or orthopaedic pathology at the cervical spine (confirmed by consultant) Have had a stroke within the last 3 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adults (over the age of 16 years) with a clinical diagnosis of neurofibromatosis 2 who attend the neurofibromatosis clinic for appointments at Guys hospital, London and who fit the inclusion/exclusion criteria for the trial are eligable to participate in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Modified nine hole peg test | Up to 3 minutes
  Participant is sitting comfortably in a chair in front of a desk. The 9 hole peg test equipment is set up so that the bowl containing pegs is directly behind the pegboard and in front of the participant. Participants can rest the forearms on the desk but must use only 1 hand for each test. If not the test is invalid. The assessor measures from the time the fingers pick up the first peg from the bowl until the fingers place the last peg in the hole of the pegboard. Time will be recorded in seconds and milliseconds.
Four square step test | Up to 30 seconds
  This is a test of balance when moving. Participants are asked to step forwards, sideways and backwards in a specific pattern. The rater times how long it takes to complete the test
Modified Clinical Test of Sensory Integration and Balance | Up to 10 minutes
  This is a test of standing balance. Participants are asked to stand upright with the feet together, first on a hard surface (the floor) and then on a soft surface (some foam). The rater will time the participant standing in each position with the eyes open and shut.

SECONDARY OUTCOMES:
Dynamic Visual Acuity test | Up to 3 minutes
  This is a test of vision when the head is turning. The participant is asked to read letters from a computer screen when the head is still then when it is being turned by a physiotherapist. The rater measures the accuracy of vision
The NFTI-QOL: A Disease-Specific Quality of Life Questionnaire for Neurofibromatosis 2 | Up to 2 minutes
  An eight question, self-report, disease specific quality of life questionnaire. Participants rate problems experienced within eight domains (balance, hearing, facial weakness, sight, walking, outlook on life, pain, mood) as no issues, slight problems, some difficulties, severe difficulties)

CONTACTS AND LOCATIONS:
Locations (1):
- Neurofibromatosis Unit, Guys Hospital., London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data with other researchers- this was not agreed in our ethical plan